CLINICAL TRIAL: NCT03300479
Title: Clevidipine (Cleviprex®) Compared With Urapidil (Ebrantil®) for Blood Pressure Reduction in Patients With Primary Intracerebral Hemorrhage: A Randomized Controlled Trial
Brief Title: Clevidipine (Cleviprex®) Compared With Urapidil (Ebrantil®)
Acronym: Clevidipine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient enrolled. No study conduct due to lack of human resources.
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Emanuela Keller, Prof. Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00379
Record Dates: First submitted 2017-09-08; First posted 2017-10-03 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Nontraumatic Intracerebral Hemorrhage, Multiple Localized
Keywords: nontraumatic intracerebral hemorrhage; Cleviprex®; Ebrantil®; Systolic blood pressure
MeSH Terms: interventions — clevidipine; urapidil

STUDY DESIGN:
Intervention Model Description: After admission to the ICU the patients presenting with primary intracerebral hemorrhage are evaluated for enrollment. If systolic blood pressure is higher than 160 mmHg or <160 mmHg under intravenous antihypertensive drug, started less than 3 h before randomizsation, the patient will be randomized in one of the two study groups and intravenous therapy with Cleviprex® or Ebrantil® will start immediately. Data of systemic haemodynamics will be collected continuously by online monitoring, starting at baseline and ending after 24h. If the target values are not attained within 30 minutes, the investigators can add or switch to alternative antihypertensive drugs of their choice. 24h after initiation of Cleviprex® or Ebrantil®, all patients receive Cardene® (standard care in daily clinical routine) for another 24h followed by orally administered antihypertensive medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clevidipine (Experimental): The treatment starts at admission to the ICU for 24 hours with 2 mg to a maximum of 16 mg Clevidipine per hour infused intravenously and continuously to reach the systolic target pressure < 160 mmHg (>120 mmHg).
  Interventions: Drug: Clevidipine
- Urapidil (Active Comparator): The treatment starts at admission to the ICU for 24 hours with 5 mg to a maximum of 40 mg Urapidil per hour infused intravenously and continuously to reach the systolic target pressure < 160 mmHg (>120 mmHg).
  Interventions: Drug: Urapidil

INTERVENTIONS:
Drug: Clevidipine — Intravenous antihypertensive therapy with Clevidipine for the first 24 hours in patients with nontraumatic intracerebral hemorrhage (ICH).
  Other Names: Cleviprex®
  Arms: Clevidipine
Drug: Urapidil — We compare the therapy with Urapidil to Clevidipine for the acute phase (24 hours) in patients with ICH. We would like to show the efficacy and safety of Clevidipine in this special situation.
  Other Names: Ebrantil®
  Arms: Urapidil

SUMMARY:
Intracerebral hemorrhage (ICH) is responsible for 10-15% of primary strokes. ICH is a dynamic process with three phases: initial hemorrhage, followed by hematoma expansion and perihematoma edema formation. Hematoma volume is correlated with disease progression and outcome. Contemporary evidence proposes that elevated blood pressure is associated with hematoma expansion while more than 90% of patients with ICH present with acute hypertension. Uncontrolled blood pressure is a leading cause of ICH and it seems also to be a factor of poorer outcomes. Therefore, rapid reduction and control of blood pressure might ease disease progression and improve the outcome. Clevidipine (Cleviprex®), an ultrashort-acting dihydropyridine calcium channel antagonist, with its rapid onset and short duration might be more effective than conventional antihypertensives to achieve rapid blood pressure control in patients with acute ICH.

DETAILED DESCRIPTION:
After admission to the ICU the patients presenting with primary intracerebral hemorrhage (ICH) are evaluated for enrollment. If systolic blood pressure (SBP) is higher than 160 mmHg or SBP <160 mmHg under intravenous antihypertensive drug (e.g. Urapidil), started less than 3 h before randomization, the patient will be randomized in one of the two study groups and intravenous therapy with Clevidipine (Cleviprex®) or Urapidil (Ebrantil®) will start immediately. Data of systemic haemodynamics will be collected continuously by online monitoring, starting at baseline and ending after 24h (study data measurements). In particular, all blood pressure measurements are extracted via an arterial line, which is placed as standard of care in these patients. If the target values are not attained within 30 minutes, the investigators can add or switch to alternative antihypertensive drugs of their choice. 24h after initiation of Clevidipine (Cleviprex®) or Urapidil (Ebrantil®), all patients receive Nicardipine (Cardene®) (standard care in daily clinical routine) for another 24h followed by orally administered antihypertensive medication.

Intracerebral hematoma volume will be determined by readings of noncontrast brain computed tomography (CT) scans using the ABC/2 rule to calculate the volume. As a standard in these patients a CT scan is performed 6 hours after admission to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Primary intracerebral hemorrhage (ICH)
* Systolic blood pressure (SBP) > 160 mmHg at screening
* Systolic blood pressure (SBP) <160 mmHg under intravenous antihypertensive drug (e.g. Urapidil), started less than 3 h before randomization
* 18 to unlimited years of age
* Signed informed consent obtained

Exclusion Criteria:

* Patients with secondary hemorrhage (bleeding source as aneurysm, arteriovenous malformation or traumatic)
* Patients with concomitant severe critical illness (e.g. sepsis, multi-organ failure)
* Positive pregnancy test for any female of childbearing potential or breast feeding female
* Known allergy to any component of Clevidipine (Cleviprex®), Urapidil Ebrantil®), soya bean oil or severe egg protein allergy
* Contraindications for Clevidipine (Cleviprex®): defect in the lipid metabolism, critical aortic stenosis
* Contraindications for Urapidil (Ebrantil®): aortic coarctation, arterio-venous shunt, breastfeeding period
* Patients with pre-existing disability and legal representative
* Patients participating in a interventional clinical trial within the last 30 days before Start of Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Achieving the target systolic blood pressure | 1/2 hours
  Number of patients achieving the target systolic blood pressure (SBP) values (160 -120 mmHg) within 30 minutes after initiation of Clevidipine (Cleviprex®) or Urapidil (Ebrantil®)

SECONDARY OUTCOMES:
Hypertensive burden - time | 24 hours
  • Hypertensive burden - time out of target range (SBP > 160 mmHg) multiplied with the numeric difference to 160mmHg
Hypotensive burden - time | 24 hours
  • Hypotensive burden - time out of target range (SBP < 120 mmHg) multiplied with the numeric difference to 120mmHg
Cumulative time out | 24 hours
  • Cumulative time out of target systolic blood pressure range (>160 or <120 mmHg)
Blood pressure variability | 48 hours
  • Blood pressure variability (determined as Standard Deviation (SD) of SBP over time)
Hematoma growth | 6 hours
  • Hematoma growth within 6 hours after admission (CCT scan)
Neurological state 1 | 48 hours
  • Glasgow Coma Scale (GCS)
Neurological state 2 | 48 hours
  • modified Ranking Scale (mRS)

OTHER OUTCOMES:
Costs | 24 hours
  • Cost of study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Keller, MD Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No